CLINICAL TRIAL: NCT06791473
Title: AI-Based Cancer Diagnosis and Prediction Using Electronic Health Records
Brief Title: AI-Driven Cancer Diagnosis and Prediction With EHR
Status: Recruiting | Type: Observational
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kang Zhang, Chief Scientist, Wenzhou Medical University
Other Study IDs: Cancer
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Tumor
Keywords: tumor; Early Disease Prediction; AI-Assisted Diagnosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Cohort: This group consists of individuals without any diagnosed cancer. Participants in this cohort will serve as the control group for comparison to the experimental group. No interventions or treatments will be administered to this cohort, as they represent a baseline of healthy individuals.
  Interventions: Diagnostic Test: AI-Based Diagnostic and Prognostic Model
- Tumor Cohort: This group consists of individuals diagnosed with cancer, including various types. Participants in this cohort will serve as the experimental group for evaluating the effectiveness of the early prediction model in identifying cancer risks and improving diagnostic accuracy.
  Interventions: Diagnostic Test: AI-Based Diagnostic and Prognostic Model

INTERVENTIONS:
Diagnostic Test: AI-Based Diagnostic and Prognostic Model — This intervention involves an AI system that integrates multimodal data, including patient medical history, laboratory test results, imaging data, and genetic information, to predict the risk of cancer. The system uses deep learning algorithms to provide real-time, accurate predictions, enabling early identification of cancer risks. By analyzing historical health data, the model aims to predict potential cancer developments, improving early detection and treatment outcomes.

SUMMARY:
This is a multi-center, clinical study designed to evaluate the application and effectiveness of an AI-assisted predictive model for identifying and diagnosing cancer, leveraging multimodal health data.

DETAILED DESCRIPTION:
Cancer diagnosis and early detection are crucial for improving patient outcomes and survival rates. Early identification of cancers and appropriate intervention can significantly impact treatment success and prognosis. In clinical practice, oncologists often need to integrate a variety of patient data-including medical history, laboratory test results, imaging data such as CT scans and MRIs, and genetic markers-to make an accurate diagnosis and develop a personalized treatment plan.

To build the foundation for our work, first phase of the project was initiated in 2023, conducting a large-scale retrospective study. This foundational phase involved analyzing comprehensive, multimodal data from approximately 1 million cancer patients. The goal was to identify key patterns and build robust preliminary models.

As precision medicine becomes increasingly important, the challenge remains to identify cancer at early stages, especially when symptoms are subtle or absent. Building on the insights from our initial analysis, the project's second phase was launched in February 2025: a prospective study. This current study aims to develop and validate an AI-assisted decision-making system by integrating multimodal data from electronic health records, imaging, laboratory results, and genetic data in a real-world clinical setting. The objective is to improve diagnostic accuracy, optimize clinical workflows, and provide more personalized treatment options for cancer patients. Ultimately, through this comprehensive, two-phase approach, this system seeks to improve early detection, guide effective treatment strategies, and enhance patient survival rates.

ELIGIBILITY:
Inclusion Criteria:

1、Patients with comprehensive electronic health records (EHRs), including medical history, laboratory test results, imaging data, and genetic data (if available).

2. Individuals without severe cognitive impairments or conditions that would prevent them from providing informed consent or participating in the study.

3. Parents or guardians must provide informed consent for minors, while adult participants must provide informed consent for themselves.

Exclusion Criteria:

1. Patients with incomplete or missing key electronic health record data or insufficient follow-up data.
2. Individuals with severe cognitive disorders or other terminal illnesses that would prevent meaningful participation.
3. Pregnant women (although pediatric cancers are being considered, pregnant women would be excluded for safety reasons).

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals aged 0 to 90 years who have received care at participating study centers. Participants must have comprehensive electronic health records (EHRs) available, including medical history, laboratory test results, imaging data, and genetic information (if available). Both individuals diagnosed with cancer (including pediatric and adult cancers) and healthy individuals with no history of cancer will be included in the study to evaluate the AI-assisted model's diagnostic and predictive capabilities. The study will focus on patients with complete and documented care records from the participating centers, ensuring a diverse cohort for analysis across different age groups and cancer types.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | 1 year
  AUC of the ROC curve, used to quantify diagnostic accuracy. No unit (a ratio or percentage, typically expressed as a number between 0 and 1).
F1 Score | 1 year
  The F1 score is the harmonic mean of precision and sensitivity (recall). It is a good measure of the model's ability to identify both true positives and minimize false positives, especially in cases where the classes are imbalanced (e.g., when the number of healthy cases is much higher than disease cases). The F1 score ranges from 0 to 1, with 1 indicating perfect precision and recall.

SECONDARY OUTCOMES:
Sensitivity (True Positive Rate) | 1 year
  Sensitivity measures how well the AI model identifies true positive cases, such as correctly diagnosing pregnant women with complications or identifying neonatal disorders.
Specificity (True Negative Rate) | 1 year
  Specificity measures the ability of the AI model to correctly identify cases without diseases, ensuring that healthy mothers and infants are correctly identified as negative.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong
  - West China Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No